CLINICAL TRIAL: NCT01343277
Title: A Randomized Controlled Study of YONDELIS (Trabectedin) or Dacarbazine for the Treatment of Advanced Liposarcoma or Leiomyosarcoma
Brief Title: A Study of Trabectedin or Dacarbazine for the Treatment of Patients With Advanced Liposarcoma or Leiomyosarcoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Collaborators: PharmaMar (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR018004; ET743SAR3007 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2011-04-26; First posted 2011-04-28 (Estimated); Results first posted 2016-01-28 (Estimated); Last update posted 2016-08-26 (Estimated); Status verified 2016-07

CONDITIONS: Advanced Liposarcoma or Leiomyosarcoma
Keywords: Advanced Liposarcoma or Leiomyosarcoma; Trabectedin; Yondelis; Dacarbazine; Anthracycline; L-sarcoma
MeSH Terms: conditions — Leiomyosarcoma | interventions — Trabectedin; Dacarbazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Trabectedin (Experimental)
  Interventions: Drug: Trabectedin
- Dacarbazine (Active Comparator)
  Interventions: Drug: Dacarbazine

INTERVENTIONS:
Drug: Trabectedin — Type=exactly number, unit=mg/m2, number=1.5, form=intravenous infusion, route=intravenous use. Once every 3 weeks until disease progression or signs of toxicity.
  Arms: Trabectedin
Drug: Dacarbazine — Type=exactly number, unit=g/m2, number=1, form=intravenous infusion, route=intravenous use. Once every 3 weeks until disease progression or signs of toxicity.
  Arms: Dacarbazine

SUMMARY:
The purpose of this study is to evaluate whether overall survival for the trabectedin group is superior to the dacarbazine group for patients with advanced L-sarcoma (liposarcoma or leiomyosarcoma).

DETAILED DESCRIPTION:
This is a randomized study (study drug assigned by chance) using a 2:1 randomization. It is an open-label (all people know study drug), active-controlled (comparing to a different drug used for the same condition), parallel-group (different treatment groups continue with separate treatments throughout the study), multicenter study. This study will be divided into 3 phases, screening, treatment, follow-up and optional extension phase (OEP). During screening, potential participants will be assessed for study eligibility after providing signed informed consent. Approximately 570 patients who satisfy all inclusion and exclusion criteria will be randomly assigned in a 2:1 ratio to either the trabectedin (n=380) or dacarbazine (n=190) treatment groups. During the treatment phase, patients will receive study drug once every 3 weeks, until disease progression (defined by Response Evaluation Criteria in Solid Tumors [RECIST] Version 1.1 criteria) or signs of toxicity. Assessments will be performed to evaluate the effectiveness of the drug, and patient safety will be monitored. During the follow-up phase, after the last dose of study drug, clinical outcomes for patients will be evaluated. Trabectedin will be administered at a dose of 1.5 milligram per square meters (mg/m^2) through a catheter into a large vein as a 24-hour intravenous (IV) infusion, once every 3 weeks, until disease progression or signs of toxicity. Dacarbazine will be administered at a dose of 1.0 g/m^2 as a 20-120 minute infusion, once every 3 weeks, until disease progression or signs of toxicity. In the OEP, participants who were previously randomized to the dacarbazine group will have the option to receive trabectedin at the discretion of the investigator.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven, unresectable, locally advanced or metastatic liposarcoma (dedifferentiated, myxoid round cell, or pleomorphic) or leiomyosarcoma. Participants must have a pathology report indicating the diagnosis of liposarcoma or leiomyosarcoma that has been reviewed by the sponsor before randomization may occur
* Treated in any order with at least: an anthracycline and ifosfamide containing regimen, or an anthracycline containing regimen and 1 additional cytotoxic chemotherapy regimen
* Measurable disease at baseline in accordance with RECIST Version 1.1
* Pathology specimens (example [e.g.], tumor blocks or unstained slides) for potential centralized pathology review and biomarker studies
* ECOG Performance Status score of 0 or 1
* Adequate recovery from prior therapy, all side effects (except alopecia) have resolved to Grade 1 or less according to the National Cancer Institute - Common Terminology Criteria of Adverse Events (NCI-CTCAE) Version 4.0
* Adequate organ function as evidenced by the following peripheral blood counts or serum chemistry values: hemoglobin 9 gram per deciliters (g/dL), absolute neutrophil count (ANC) 1,500/L, platelet count 100,000/L, serum creatinine 1.5*the upper limit of normal (ULN), creatine phosphokinase (CPK) 2.5 Upper Limit of Normal [ULN]
* Adequate hepatic function as evidenced by the following serum chemistry values: total bilirubin, ULN. If total bilirubin is greater than (>) ULN, measure indirect bilirubin to evaluate for Gilbert's syndrome (if direct bilirubin is within normal range, participant may be eligible) ALP 2.5 x ULN; Trabectedin: if the ALP is >2.5 x ULN, then an ALP liver fraction or 5-nucleotidase must be obtained and ULN, AST and ALT 2.5 ULN
* Negative pregnancy test (urinary or serum beta-HCG) at screening (applicable to women of child bearing potential who are sexually active)
* Female participants must be postmenopausal (no spontaneous menses for at least 2 years), surgically sterile (have had a hysterectomy or bilateral oophorectomy, tubal ligation, or otherwise be incapable of pregnancy), abstinent (at the discretion of the investigator), or if sexually active, be practicing an effective method of birth control. Male participants must agree to use an adequate contraception method as deemed appropriate by the investigator (e.g., vasectomy, double-barrier, partner using effective contraception) and to not donate sperm for a minimum of 5 months after treatment discontinuation

Optional Extension Phase (OEP) Phase:

* Documentation for inclusion criteria histologically proven, unresectable, locally advanced or metastatic liposarcoma (dedifferentiated, myxoid round cell, or pleomorphic) or leiomyosarcoma. Participants must have a pathology report indicating the diagnosis of liposarcoma or leiomyosarcoma that has been reviewed by the sponsor before randomization may occur and treated in any order with at least: an anthracycline and ifosfamide containing regimen, or an anthracycline containing regimen and 1 additional cytotoxic chemotherapy regimen do not need to be reviewed by the Sponsor
* Collection of the specimen: Pathology specimens (example (e.g.), tumor blocks or unstained slides) for potential centralized pathology review and biomarker studies is not applicable
* Documentation of inclusion criteria adequate organ function as evidenced by the following peripheral blood counts or serum chemistry values: hemoglobin 9 gram per deciliters (g/dL), absolute neutrophil count (ANC) 1,500/L, platelet count 100,000/L, serum creatinine 1.5*the upper limit of normal (ULN), creatine phosphokinase (CPK) 2.5*ULN and adequate hepatic function as evidenced by the following serum chemistry values: total bilirubin, ULN. If total bilirubin is greater than (>) ULN, measure indirect bilirubin to evaluate for Gilbert's syndrome (if direct bilirubin is within normal range, participant may be eligible) ALP <= 2.5*ULN; Trabectedin: if the ALP is >2.5*ULN, then an ALP liver fraction or 5-nucleotidase must be obtained and ULN, AST and ALT 2.5 ULN will be reviewed by the Sponsor before enrollment in the OEP may occur

Exclusion Criteria:

* Potential participants who meet any of the following criteria will be excluded from participating in the study: Prior exposure to trabectedin or dacarabazine, less than 3 weeks from last dose of systemic cytotoxic therapy, radiation therapy, or therapy with any investigational agent, other malignancy within past 3 years. Exceptions: basal or nonmetastatic squamous cell carcinoma of the skin, cervical carcinoma in situ, or Federation Internationale de Gynecologie et d'Obstetrique (FIGO) Stage 1 carcinoma of the cervix
* Known central nervous system metastasis
* Known significant chronic liver disease, such as cirrhosis or active hepatitis (potential participants who test positive for hepatitis B surface antigen or hepatitis C antibodies are allowed provided they do not have active disease requiring antiviral therapy)
* Myocardial infarct within 6 months before enrollment, New York Heart Association Class II or greater heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, clinically significant pericardial disease, or electrocardiographic evidence of acute ischemic or active conduction system abnormalities
* Uncontrolled intercurrent illness including, but not limited to, poorly controlled hypertension or diabetes, ongoing active infection, or psychiatric illness/social situation that may potentially impair the participant's compliance with study procedures
* Unwilling or unable to have a central venous catheter
* Known allergies, hypersensitivity, or intolerance to trabectedin, dacarbazine, dexamethasone, or their excipients
* Pregnant or breast-feeding
* Any condition that, in the opinion of the investigator, would compromise the well-being of the participant or the study or prevent the participant from meeting or performing study requirements

OEP phase:

* Potential participants who meet any of the following criteria will be excluded from Participating in the study: Prior exposure to trabectedin, less than 3 weeks from last dose of systemic cytotoxic therapy, radiation therapy, or therapy with any investigational agent, other malignancy within past 3 years. Exceptions: basal or nonmetastatic squamous cell carcinoma of the skin, cervical carcinoma in situ, or Federation Internationale de Gynecologie et d'Obstetrique (FIGO) Stage 1 carcinoma of the cervix does not apply
* Treated in any order with at least: an anthracycline and ifosfamide containing regimen, or an anthracycline containing regimen and 1 additional cytotoxic chemotherapy regimen with less than 3 weeks from last dose of systemic anticancer therapy, radiation therapy, or therapy with any investigational agent
* Known allergies, hypersensitivity, or intolerance to dacarbazine does not apply

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 579 (Actual)
Dates: Start 2011-06; Primary Completion 2015-01 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (88):
- United States (77):
  - Phoenix, Arizona
  - Tucson, Arizona
  - Little Rock, Arkansas
  - La Jolla, California
  - Los Angeles, California
  - San Diego, California
  - San Francisco, California
  - Santa Monica, California
  - Aurora, Colorado
  - Denver, Colorado
  - Hartford, Connecticut
  - New Haven, Connecticut
  - Boynton Beach, Florida
  - Hollywood, Florida
  - Miami, Florida
  - Orlando, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Augusta, Georgia
  - Savannah, Georgia
  - Post Falls, Idaho
  - Chicago, Illinois
  - Naperville, Illinois
  - Park Ridge, Illinois
  - Peoria, Illinois
  - Springfield, Illinois
  - Indianapolis, Indiana
  - Iowa City, Iowa
  - Sioux City, Iowa
  - Overland Park, Kansas
  - Wichita, Kansas
  - Louisville, Kentucky
  - Covington, Louisiana
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Ann Arbor, Michigan
  - Detroit, Michigan
  - Lansing, Michigan
  - Jackson, Mississippi
  - Saint Joseph, Missouri
  - St Louis, Missouri
  - Omaha, Nebraska
  - Henderson, Nevada
  - Las Vegas, Nevada
  - Lebanon, New Hampshire
  - Hackensack, New Jersey
  - Morristown, New Jersey
  - Newark, New Jersey
  - Albuquerque, New Mexico
  - Johnson City, New York
  - New York, New York
  - Syracuse, New York
  - The Bronx, New York
  - Chapel Hill, North Carolina
  - Charlotte, North Carolina
  - Akron, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Oklahoma City, Oklahoma
  - Tulsa, Oklahoma
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - State College, Pennsylvania
  - Charleston, South Carolina
  - Knoxville, Tennessee
  - Nashville, Tennessee
  - Austin, Texas
  - Dallas, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Fairfax, Virginia
  - Seattle, Washington
  - Morgantown, West Virginia
  - Green Bay, Wisconsin
  - Milwaukee, Wisconsin
- Australia (4):
  - Malvern
  - Randwick
  - Subiaco
  - Woolloongabba
- Brazil (5):
  - Bahia
  - Barretos
  - Ijuí
  - Porto Alegre
  - São Paulo
- New Zealand (2):
  - Auckland
  - Wellington

REFERENCES:
- [Derived] Jones RL, Herzog TJ, Patel SR, von Mehren M, Schuetze SM, Van Tine BA, Coleman RL, Knoblauch R, Triantos S, Hu P, Shalaby W, McGowan T, Monk BJ, Demetri GD. Cardiac safety of trabectedin monotherapy or in combination with pegylated liposomal doxorubicin in patients with sarcomas and ovarian cancer. Cancer Med. 2021 Jun;10(11):3565-3574. doi: 10.1002/cam4.3903. Epub 2021 May 7. PMID 33960681
- [Derived] Patel S, von Mehren M, Reed DR, Kaiser P, Charlson J, Ryan CW, Rushing D, Livingston M, Singh A, Seth R, Forscher C, D'Amato G, Chawla SP, McCarthy S, Wang G, Parekh T, Knoblauch R, Hensley ML, Maki RG, Demetri GD. Overall survival and histology-specific subgroup analyses from a phase 3, randomized controlled study of trabectedin or dacarbazine in patients with advanced liposarcoma or leiomyosarcoma. Cancer. 2019 Aug 1;125(15):2610-2620. doi: 10.1002/cncr.32117. Epub 2019 Jun 7. PMID 31173362
- [Derived] Jones RL, Demetri GD, Schuetze SM, Milhem M, Elias A, Van Tine BA, Hamm J, McCarthy S, Wang G, Parekh T, Knoblauch R, Hensley ML, Maki RG, Patel S, von Mehren M. Efficacy and tolerability of trabectedin in elderly patients with sarcoma: subgroup analysis from a phase III, randomized controlled study of trabectedin or dacarbazine in patients with advanced liposarcoma or leiomyosarcoma. Ann Oncol. 2018 Sep 1;29(9):1995-2002. doi: 10.1093/annonc/mdy253. PMID 30084934
- [Derived] Calvo E, Azaro A, Rodon J, Dirix L, Huizing M, Senecal FM, LoRusso P, Yee L, Poggesi I, de Jong J, Triantos S, Park YC, Knoblauch RE, Parekh TV, Demetri GD, von Mehren M. Hepatic safety analysis of trabectedin: results of a pharmacokinetic study with trabectedin in patients with hepatic impairment and experience from a phase 3 clinical trial. Invest New Drugs. 2018 Jun;36(3):476-486. doi: 10.1007/s10637-017-0546-9. Epub 2017 Nov 27. PMID 29177975
- [Derived] Demetri GD, von Mehren M, Jones RL, Hensley ML, Schuetze SM, Staddon A, Milhem M, Elias A, Ganjoo K, Tawbi H, Van Tine BA, Spira A, Dean A, Khokhar NZ, Park YC, Knoblauch RE, Parekh TV, Maki RG, Patel SR. Efficacy and Safety of Trabectedin or Dacarbazine for Metastatic Liposarcoma or Leiomyosarcoma After Failure of Conventional Chemotherapy: Results of a Phase III Randomized Multicenter Clinical Trial. J Clin Oncol. 2016 Mar 10;34(8):786-93. doi: 10.1200/JCO.2015.62.4734. Epub 2015 Sep 14. PMID 26371143

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Total enrolled participants were 577, but 2 participants were randomized twice, therefore counted twice in enrollment. Thus, enrolled participants are reported as 579.
Groups:
- Trabectedin: Trabectedin at a dose of 1.5 milligram per meter square (mg/m^2) was given as an intravenous (IV) infusion over 24-hour every 3 weeks on Day 1 of every cycle (21 days) until disease progression. Dexamethasone 20 mg IV was also administered within 30 minutes before start of each trabectedin infusion.
- Dacarbazine: Dacarbazine at a dose of 1 gram per meter square (mg/m^2) was given as an intravenous (IV) infusion over 20-120 minutes every 3 weeks on Day 1 of every cycle (21 days) until disease progression. Dexamethasone 20 mg IV was also administered within 30 minutes before start of each dacarbazine infusion.
Period: Overall Study
Arm/Group | Trabectedin | Dacarbazine
Started | 384 | 193
Treated | 378 | 172
Completed | 0 | 0
Not Completed | 384 | 193
Not completed — Other | 3 | 3
Not completed — Withdrawal by Subject | 18 | 13
Not completed — Physician Decision | 1 | 2
Not completed — Death | 10 | 1
Not completed — Adverse Event | 67 | 13
Not completed — Disease progression | 270 | 138
Not completed — Randomized not treated | 6 | 21
Not completed — Treatment ongoing | 8 | 2
Not completed — Subsequent anticancer therapy | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Trabectedin | Dacarbazine | Total
Number analyzed (Participants) | 384 | 193 | 577
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.5 (11.04) | 54.1 (11.92) | 55.7 (11.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 262 | 140 | 402
  Male | 122 | 53 | 175
Region of Enrollment [Number; unit: participants]
  AUS | 15 | 8 | 23
  BRA | 10 | 2 | 12
  NZL | 3 | 0 | 3
  USA | 356 | 183 | 539

OUTCOME MEASURES:

1. Secondary Outcome: Progression-Free Survival (PFS)
Description: The Progression-Free Survival (PFS) was assessed as median number of months from baseline until the first documented sign of disease progression (increase in disease; radiographic, clinical, or both) or death due to any cause, whichever occurred earlier. Independent Data Monitoring Committee performed ongoing safety monitoring and conducted the interim analysis after 189 death events and 329 PFS events were observed.
Time Frame: approximately 2 years 4 months (From Study start date [27 May 2011] up to interim analysis data cut-off [16 September 2013])
Population: Analysis population included all the randomized participants up to interim analysis cut-off date (16 September 2013). "N" (number of participants analyzed) signifies the participants evaluable for this measure.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Trabectedin | Dacarbazine
Number analyzed (Participants) | 345 | 173
Months | 4.21 [2.99 to 4.83] | 1.54 [1.48 to 2.60]

2. Secondary Outcome: Time to Progression
Description: Time interval in months between the date of randomization and the date of disease progression or death due to progression, whichever occurred first.
  Independent Data Monitoring Committee performed ongoing safety monitoring and conducted the interim analysis after 189 death events and 329 PFS events were observed.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Trabectedin | Dacarbazine
Number analyzed (Participants) | 345 | 173
Months | 4.24 [3.22 to 4.93] | 1.54 [1.48 to 2.60]

3. Secondary Outcome: Objective Response Rate
Description: The objective response rate (ORR) is defined as the percentage of participants who achieved a Complete response (CR) or partial response (PR) as best responses. according to Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST). CR defined as disappearance of all target lesions. Any pathological lymph nodes must have reduction in short axis to less than 10 millimeter (mm). PR defined as at least 30 percent (%) decrease in sum of the diameters of the target lesions taking as reference the Baseline sum diameters. Confirmed responses are those that persist on repeat imaging study for at least 4 weeks after initial documentation of response. Independent Data Monitoring Committee performed ongoing safety monitoring and conducted the interim analysis after 189 death events and 329 PFS events were observed.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Trabectedin | Dacarbazine
Number analyzed (Participants) | 345 | 173
Percentage of Participants | 9.9 [6.9 to 13.5] | 6.9 [3.6 to 11.8]

4. Secondary Outcome: Duration of Response
Description: Duration of response is defined as the time from the date of initial documentation of a response (CR or PR) to the date of first documented evidence of progressive disease (or relapse for participants who experience CR during the study) or death.
  Independent Data Monitoring Committee performed ongoing safety monitoring and conducted the interim analysis after 189 death events and 329 PFS events were observed.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Trabectedin | Dacarbazine
Number analyzed (Participants) | 34 | 12
Months | 6.47 [3.58 to 7.62] | 4.17 [2.14 to NA] — Insufficient participants reached the median percentile to calculate the upper limits of confidence interval.

5. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: approximately 3 years 8 months (From Study start date [27 May 2011] up to final analysis data cut-off [05 January 2015])
Population: Safety population included all the treated participants.
Measure: Number; unit: Participants
Arm/Group | Trabectedin | Dacarbazine
Number analyzed (Participants) | 378 | 172
Participants
  Serious Adverse Events (SAEs) | 155 | 52
  Adverse Events (AEs) | 375 | 166

6. Primary Outcome: Overall Survival (OS)
Description: The OS is defined as the time from the date of first dose of study drug to date of death from any cause. If the participant is alive or the vital status is unknown, the participant will be censored at the date the participant will be last known to be alive.
Time Frame: approximately 3 years 8 months (From Study start date [27 May 2011] up to final analysis data cut-off [05 January 2015]
Population: Analysis population included all the randomized participants up to up to final analysis cut-off date (05 January 2015).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Trabectedin | Dacarbazine
Number analyzed (Participants) | 384 | 193
Months | 13.73 [12.16 to 16.00] | 13.14 [9.10 to 16.23]

ADVERSE EVENTS:
Time Frame: approximately 3 years 8 months (From Study start date [27 May 2011] up to final analysis data cut-off [05 January 2015]
Description: Safety population included all the treated participants.
Arm/Group | Trabectedin | Dacarbazine
Serious Adverse Events (participants affected / at risk) | 155/378 | 52/172
Other Adverse Events (participants affected / at risk) | 375/378 | 166/172
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Trabectedin (N=378) | Dacarbazine (N=172)
Anaemia (Blood and lymphatic system disorders) | 15 | 4
Febrile Neutropenia (Blood and lymphatic system disorders) | 12 | 2
Leukocytosis (Blood and lymphatic system disorders) | 3 | 0
Leukopenia (Blood and lymphatic system disorders) | 4 | 3
Microangiopathic Haemolytic Anaemia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 9 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 7 | 3
Atrial Fibrillation (Cardiac disorders) | 2 | 1
Atrial Flutter (Cardiac disorders) | 1 | 0
Cardiac Arrest (Cardiac disorders) | 3 | 0
Cardiac Disorder (Cardiac disorders) | 1 | 0
Cardiac Failure (Cardiac disorders) | 3 | 0
Cardiac Failure Acute (Cardiac disorders) | 1 | 0
Cardiac Failure Congestive (Cardiac disorders) | 7 | 0
Cardiomyopathy (Cardiac disorders) | 2 | 0
Left Ventricular Dysfunction (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0
Right Ventricular Dysfunction (Cardiac disorders) | 1 | 0
Sinus Tachycardia (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0
Visual Impairment (Eye disorders) | 1 | 0
Abdominal Distension (Gastrointestinal disorders) | 0 | 1
Abdominal Hernia (Gastrointestinal disorders) | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 13 | 8
Abdominal Pain Lower (Gastrointestinal disorders) | 2 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 2 | 0
Colitis (Gastrointestinal disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 4 | 0
Duodenal Obstruction (Gastrointestinal disorders) | 1 | 2
Dysphagia (Gastrointestinal disorders) | 2 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 2 | 0
Intestinal Obstruction (Gastrointestinal disorders) | 3 | 0
Intestinal Ulcer (Gastrointestinal disorders) | 0 | 1
Intra-Abdominal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Large Intestinal Obstruction (Gastrointestinal disorders) | 0 | 1
Large Intestine Perforation (Gastrointestinal disorders) | 1 | 0
Lower Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 15 | 3
Obstruction Gastric (Gastrointestinal disorders) | 1 | 1
Oesophageal Obstruction (Gastrointestinal disorders) | 1 | 0
Oesophageal Pain (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 3 | 0
Rectal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 9 | 3
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 15 | 3
Asthenia (General disorders) | 5 | 0
Catheter Site Inflammation (General disorders) | 1 | 0
Chest Discomfort (General disorders) | 1 | 0
Chest Pain (General disorders) | 1 | 0
Death (General disorders) | 5 | 3
Device Breakage (General disorders) | 1 | 0
Device Failure (General disorders) | 1 | 0
Fatigue (General disorders) | 4 | 1
Gait Disturbance (General disorders) | 1 | 0
Generalised Oedema (General disorders) | 1 | 0
Infusion Site Extravasation (General disorders) | 2 | 0
Malaise (General disorders) | 1 | 0
Multi-Organ Failure (General disorders) | 1 | 0
Necrosis (General disorders) | 1 | 0
Non-Cardiac Chest Pain (General disorders) | 0 | 1
Oedema Peripheral (General disorders) | 2 | 1
Pain (General disorders) | 1 | 1
Pyrexia (General disorders) | 12 | 2
Thrombosis in Device (General disorders) | 1 | 0
Hepatotoxicity (Hepatobiliary disorders) | 1 | 0
Portal Vein Thrombosis (Hepatobiliary disorders) | 1 | 0
Drug Hypersensitivity (Immune system disorders) | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1
Bacteraemia (Infections and infestations) | 2 | 0
Catheter Site Infection (Infections and infestations) | 8 | 1
Cellulitis (Infections and infestations) | 2 | 0
Clostridium Difficile Colitis (Infections and infestations) | 1 | 0
Clostridium Difficile Infection (Infections and infestations) | 1 | 0
Clostridium Difficile Sepsis (Infections and infestations) | 1 | 0
Enterococcal Bacteraemia (Infections and infestations) | 1 | 0
Kidney Infection (Infections and infestations) | 1 | 0
Lobar Pneumonia (Infections and infestations) | 1 | 0
Lung Infection (Infections and infestations) | 2 | 0
Osteomyelitis (Infections and infestations) | 0 | 1
Peritonitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 6 | 0
Respiratory Tract Infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 8 | 0
Septic Shock (Infections and infestations) | 2 | 0
Staphylococcal Bacteraemia (Infections and infestations) | 1 | 0
Urinary Tract Infection (Infections and infestations) | 7 | 2
Urinary Tract Infection Staphylococcal (Infections and infestations) | 1 | 0
Vaginal Infection (Infections and infestations) | 1 | 0
Wound Abscess (Infections and infestations) | 1 | 0
Ankle Fracture (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 0
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Vascular Access Complication (Injury, poisoning and procedural complications) | 1 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 0
Alanine Aminotransferase Increased (Investigations) | 2 | 0
Aspartate Aminotransferase Increased (Investigations) | 3 | 0
Blood Bilirubin Increased (Investigations) | 0 | 1
Blood Creatine Phosphokinase Increased (Investigations) | 4 | 0
Blood Creatinine Increased (Investigations) | 4 | 0
Blood Lactic Acid Increased (Investigations) | 0 | 1
Ejection Fraction Decreased (Investigations) | 5 | 0
International Normalised Ratio Increased (Investigations) | 2 | 0
Liver Function Test Abnormal (Investigations) | 2 | 0
Myoglobin Blood Increased (Investigations) | 1 | 0
Neutrophil Count Decreased (Investigations) | 4 | 1
Platelet Count Decreased (Investigations) | 4 | 2
Transaminases Increased (Investigations) | 2 | 0
Troponin I Increased (Investigations) | 2 | 0
White Blood Cell Count Decreased (Investigations) | 2 | 0
Acidosis (Metabolism and nutrition disorders) | 1 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 3 | 1
Dehydration (Metabolism and nutrition disorders) | 15 | 3
Failure to Thrive (Metabolism and nutrition disorders) | 2 | 0
Fluid Overload (Metabolism and nutrition disorders) | 1 | 0
Fluid Retention (Metabolism and nutrition disorders) | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 0
Hyperlipasaemia (Metabolism and nutrition disorders) | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1
Malnutrition (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 3 | 2
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint Range of Motion Decreased (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint Swelling (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 2 | 2
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 4 | 0
Soft Tissue Necrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Cancer Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Malignant Ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Cerebrovascular Accident (Nervous system disorders) | 2 | 0
Dizziness (Nervous system disorders) | 1 | 0
Haemorrhage Intracranial (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Neuralgia (Nervous system disorders) | 0 | 2
Pyramidal Tract Syndrome (Nervous system disorders) | 0 | 1
Spinal Cord Compression (Nervous system disorders) | 1 | 2
Syncope (Nervous system disorders) | 3 | 2
Confusional State (Psychiatric disorders) | 3 | 0
Mental Status Changes (Psychiatric disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 1
Obstructive Uropathy (Renal and urinary disorders) | 1 | 0
Renal Failure (Renal and urinary disorders) | 1 | 0
Renal Failure Acute (Renal and urinary disorders) | 12 | 1
Renal Tubular Necrosis (Renal and urinary disorders) | 1 | 0
Urinary Retention (Renal and urinary disorders) | 2 | 0
Urinary Tract Obstruction (Renal and urinary disorders) | 1 | 0
Pelvic Pain (Reproductive system and breast disorders) | 2 | 0
Perineal Fistula (Reproductive system and breast disorders) | 1 | 0
Vaginal Haemorrhage (Reproductive system and breast disorders) | 0 | 1
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchial Obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 13 | 2
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 6 | 1
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Respiratory Arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 6 | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hip Surgery (Surgical and medical procedures) | 1 | 0
Circulatory Collapse (Vascular disorders) | 0 | 1
Deep Vein Thrombosis (Vascular disorders) | 3 | 1
Embolism (Vascular disorders) | 1 | 0
Embolism Venous (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 4 | 1
Jugular Vein Thrombosis (Vascular disorders) | 1 | 0
Temporal Arteritis (Vascular disorders) | 0 | 1
Venous Thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Trabectedin (N=378) | Dacarbazine (N=172)
Anaemia (Blood and lymphatic system disorders) | 149 | 48
Leukopenia (Blood and lymphatic system disorders) | 43 | 11
Neutropenia (Blood and lymphatic system disorders) | 111 | 31
Thrombocytopenia (Blood and lymphatic system disorders) | 70 | 33
Abdominal Distension (Gastrointestinal disorders) | 30 | 16
Abdominal Pain (Gastrointestinal disorders) | 58 | 29
Abdominal Pain Upper (Gastrointestinal disorders) | 19 | 8
Constipation (Gastrointestinal disorders) | 140 | 52
Diarrhoea (Gastrointestinal disorders) | 130 | 40
Dry Mouth (Gastrointestinal disorders) | 22 | 13
Dyspepsia (Gastrointestinal disorders) | 30 | 12
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 12 | 11
Nausea (Gastrointestinal disorders) | 282 | 85
Stomatitis (Gastrointestinal disorders) | 21 | 6
Vomiting (Gastrointestinal disorders) | 167 | 35
Catheter Site Pain (General disorders) | 19 | 1
Chest Pain (General disorders) | 19 | 6
Chills (General disorders) | 34 | 11
Fatigue (General disorders) | 260 | 90
Influenza Like Illness (General disorders) | 19 | 6
Oedema Peripheral (General disorders) | 107 | 21
Pain (General disorders) | 18 | 9
Pyrexia (General disorders) | 64 | 27
Upper Respiratory Tract Infection (Infections and infestations) | 24 | 10
Urinary Tract Infection (Infections and infestations) | 29 | 8
Alanine Aminotransferase Increased (Investigations) | 186 | 12
Aspartate Aminotransferase Increased (Investigations) | 141 | 10
Blood Alkaline Phosphatase Increased (Investigations) | 87 | 16
Blood Bilirubin Increased (Investigations) | 34 | 5
Blood Creatine Phosphokinase Increased (Investigations) | 54 | 2
Blood Creatinine Increased (Investigations) | 47 | 3
Lymphocyte Count Decreased (Investigations) | 21 | 4
Neutrophil Count Decreased (Investigations) | 93 | 24
Platelet Count Decreased (Investigations) | 61 | 29
Weight Decreased (Investigations) | 27 | 5
White Blood Cell Count Decreased (Investigations) | 96 | 20
Decreased Appetite (Metabolism and nutrition disorders) | 138 | 36
Dehydration (Metabolism and nutrition disorders) | 43 | 17
Hyperglycaemia (Metabolism and nutrition disorders) | 30 | 5
Hypoalbuminaemia (Metabolism and nutrition disorders) | 32 | 7
Hypocalcaemia (Metabolism and nutrition disorders) | 27 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 53 | 22
Hyponatraemia (Metabolism and nutrition disorders) | 26 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 57 | 15
Back Pain (Musculoskeletal and connective tissue disorders) | 65 | 28
Bone Pain (Musculoskeletal and connective tissue disorders) | 20 | 12
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 25 | 4
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 29 | 14
Myalgia (Musculoskeletal and connective tissue disorders) | 47 | 11
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 47 | 15
Dizziness (Nervous system disorders) | 46 | 21
Dysgeusia (Nervous system disorders) | 34 | 11
Headache (Nervous system disorders) | 94 | 33
Hypoaesthesia (Nervous system disorders) | 22 | 3
Paraesthesia (Nervous system disorders) | 22 | 9
Anxiety (Psychiatric disorders) | 40 | 13
Depression (Psychiatric disorders) | 30 | 7
Insomnia (Psychiatric disorders) | 55 | 16
Cough (Respiratory, thoracic and mediastinal disorders) | 85 | 36
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 91 | 33
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 26 | 4
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 23 | 6
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 19 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 13 | 9
Flushing (Vascular disorders) | 19 | 9
Hot Flush (Vascular disorders) | 13 | 10
Hypertension (Vascular disorders) | 22 | 2
Hypotension (Vascular disorders) | 19 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.